CLINICAL TRIAL: NCT02627638
Title: Cancer Patient Perceptions of the Osteopathy Treatment: a Qualitative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013.826
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2015-09

CONDITIONS: Cancer Patients
Keywords: osteopathy; complementary therapy; symptoms in cancer patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Osteopathic treatment (Other)
  Interventions: Other: Ostheopathic treatment

INTERVENTIONS:
Other: Ostheopathic treatment — Once their clinical data were collected and their symptoms were assessed, all the enrolled patients had an osteopathic session a week during two weeks. After those sessions, they had an interview (scheduled between D11 and D14) with a psychologist

SUMMARY:
For more than seven years an osteopath has been working in the palliative care unit (PCU) and in both palliative care mobile team (PCMT) as a member of the multidisciplinary team. The patients referred to the osteopath by the palliative care physicians present pains related to cancer, but also to the treatment, in particular to surgery or radiotherapy. The osteopath can help with other symptoms such as constipation or dyspnoea. As this approach is provided in complement of the medicinal approach, it is not considered as an alternative medicine but as a complementary medicine associated to a conventional care. It seemed relevant to the investigators to ask the cancer patients undergoing osteopathic sessions for pain how they saw this complementary therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced illness patients with cancer pain, PS 0 to 2, willing to take part in the study and having signed the informed consent form

Exclusion Criteria:

* Non-communicating patients and patients whose cancer has been cured.
* Patients with fractural risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Thoughs and emotions of patients undergoing the two osteopathic sessions as complementary therapy for pain, evaluated using semi-directed interviews | around day 14 (after the second session)
  Once clinical data were collected and symptoms were assessed, all the enrolled patients had an osteopathic session a week during two weeks. After those sessions, they had an interview (scheduled between J11 and J14) with a psychologist. The research assistant psychologist conducted the semi-directed interviews. The interview questions were geared toward eliciting open-ended responses to acquire specific information about the patient thoughts and emotions associated with osteopathic treatment. In our study, we conducted two preliminary interviews to test the quality of the questions we planned to use with the participants. The specific questions that were used during the interview are available on request from the authors.

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine palliative - Groupement Hospitalier Lyon Sud- Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Result] Steel A, Tricou C, Monsarrat T, Ruer M, Deslandes C, Sisoix C, Filbet M. The perceptions and experiences of osteopathic treatment among cancer patients in palliative care: a qualitative study. Support Care Cancer. 2018 Oct;26(10):3627-3633. doi: 10.1007/s00520-018-4233-y. Epub 2018 May 4. PMID 29728845